CLINICAL TRIAL: NCT04278118
Title: HiPPI: A Phase 2 Trial of Hypofractionated Pencil Beam Scanning Proton Therapy for Benign Intracranial Tumors
Brief Title: Hypofractionated Proton Therapy for Benign Intracranial Brain Tumors, the HiPPI Study
Acronym: HiPPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bree Eaton, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00114529; NCI-2019-06446 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD4811-19 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-20 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Grade I Meningioma; Grade II Meningioma; Grade III Meningioma; Intracranial Neoplasm; Nerve Sheath Neoplasm; Pituitary Gland Adenoma; Schwannoma
MeSH Terms: conditions — Meningioma; Brain Neoplasms; Nerve Sheath Neoplasms; Pituitary Neoplasms; Neurilemmoma | interventions — Radiation Dose Hypofractionation; Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (hypofractionated radiation therapy) (Experimental): Patients with benign and radiographically diagnosed intracranial tumors undergo hypofractionated proton or photon radiation therapy daily, Monday-Friday over 17 fractions for 3.5-4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Radiation: Photon Beam Radiation Therapy; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Cohort II (hypofractionated radiation therapy) (Experimental): Patients with pathologically confirmed World Health Organization (WHO) grade 2-3 meningiomas undergo hypofractionated proton or photon radiation therapy daily, Monday-Friday over 20 fractions for 3.5-4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Radiation: Photon Beam Radiation Therapy; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated proton or photon radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation
Radiation: Photon Beam Radiation Therapy — Undergo hypofractionated proton or photon radiation therapy
Radiation: Proton Beam Radiation Therapy — Undergo hypofractionated proton or photon radiation therapy
  Other Names: PBRT; Proton Radiation Therapy; Radiation, Proton Beam
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well hypofractionated proton or photon radiation therapy works in treating patients with brain tumors. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells. A shorter duration of radiation treatment may avoid some of the delayed side effects of radiation while providing a more convenient treatment and reducing costs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To report 3 year local tumor control of moderately hypofractionated proton or photon therapy for benign intracranial tumors.

SECONDARY OBJECTIVES:

I. To demonstrate feasibility of moderate hypofractionation pencil beam scanning proton therapy for intracranial tumors.

II. To report physician reported acute and late toxicity of moderate hypofractionation pencil beam scanning proton therapy for intracranial tumors according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

III. To report neurocognitive effects, health related quality of life, and patient reported toxicity for moderate hypofractionation pencil beam scanning proton therapy for intracranial tumors.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients with benign and radiographically diagnosed intracranial tumors undergo hypofractionated proton or photon radiation therapy daily, Monday-Friday over 17 fractions for 3.5-4 weeks in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients with pathologically confirmed World Health Organization (WHO) grade 2-3 meningiomas undergo hypofractionated proton or photon radiation therapy daily, Monday-Friday over 20 fractions for 3.5-4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or radiographically diagnosed benign intracranial or nerve sheath tumor, including meningiomas, pituitary adenomas, schwannomas. World Health Organization (WHO) grade 2-3 meningiomas are also allowed
* Recommended to receive proton or photon fractionated radiation therapy
* Signed informed consent

Exclusion Criteria:

* Pregnant females are excluded. Female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy. FCBP must agree to use adequate contraception (at least one highly effective method and one additional method of birth control at the same time or complete abstinence) prior to study entry, for the duration of study. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.

  * A female of childbearing potential (FCBP) is a sexually mature woman who: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (if age >= 55 years); if the female subject is < 55 years and she has been naturally postmenopausal for >= 1 year her reproductive status has to be verified by additional laboratory (lab) tests (< 20 estradiol OR estradiol < 40 with follicle stimulating hormone [FSH] > 40 in women not on estrogen replacement therapy)
* Prior radiation therapy that would overlap with current target volume
* Inability to undergo magnetic resonance imaging (MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
local tumor control | Up to 3 years since enrollment
  Will assess local tumor control rate. Local tumor control is defined as freedom from progressive disease (PD). Will be calculated as the proportion of patients who did not experience PD within 3-year follow up with 95% binomial proportion confidence interval for the entire population and each cohort independently. The same calculation will be repeated for the entire study population and each cohort separately. Kaplan-Meier method will be used to estimate the local control rates for the entire population and each cohort independently.
Incidence of adverse events | up to 3 years
  Will be assessed and graded according to Common Terminology Criteria for Adverse Events version 5.0

SECONDARY OUTCOMES:
Neurocognitive effects | Up to 3 years
  Will be summarized by summary statistics.
Health related quality of life | Up to 3 years
  Will be summarized by summary statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Bree R Eaton, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided